CLINICAL TRIAL: NCT06206187
Title: ICE Detector-RCT: Blinded, Randomized Controlled Trial of Electrophysiologist vs. Artificial Intelligence Detection of Intracardiac Thrombus
Brief Title: Blinded Randomized Controlled Trial of Artificial Intelligence Guided Detection of Intracardiac Thrombus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Xu Liu, professor, Shanghai Chest Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ICE Detector-RCT
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrophysiologist judgment (Active Comparator)
  Interventions: Other: Electrophysiologist judgment of the intracardiac thrombus
- Artificial Intelligence Detection (Experimental)
  Interventions: Other: Automated detection of the intracardiac thrombus through deep learning

INTERVENTIONS:
Other: Automated detection of the intracardiac thrombus through deep learning — A deep learning model will identify the intracardiac thrombus. The AI model will produce an assessment of intracardiac thrombus using video based features.
  Arms: Artificial Intelligence Detection
Other: Electrophysiologist judgment of the intracardiac thrombus — Cardiac electrophysiologists use their own experience to determine whether there is intracardiac thrombus
  Arms: Electrophysiologist judgment

SUMMARY:
To determine whether an integrated AI decision support can save time and improve the accuracy of detection of intracardiac thrombus, the investigators are conducting a blinded, randomized controlled study of AI-guided detection of intracardiac thrombus to electrophysiologist judgment in preliminary readings of echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years.
2. Willing to sign informed consent.
3. Patients diagnosed with atrial fibrillation Paroxysmal AF and Persistent AF according to the latest clinical guidelines

Exclusion Criteria:

1. End-stage disease with a mean life expectancy less than 1 year
2. New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction less than 30%
3. Previous surgical or catheter ablation for AF
4. Bradycardia and presence of implanted ICD
5. Uncontrolled hypertension: Systolic blood pressure (SBP) >180 mmHg or diastolic blood pressure (DBP) > 110 mmHg
6. Patients with Cardiovascular events including acute myocardial infarction, any PCI, valvular cardiac surgical, or percutaneous procedure within the past 3 months
7. Women of childbearing potential who are, or plan to become, pregnant during the time of the study
8. Have been enrolled in an investigational study evaluating devices or drugs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2024-01-05 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of change from initial (AI vs EP doctor) assessment to final cardiologist assessment | 10 Minutes

SECONDARY OUTCOMES:
Perioperative adverse event rates | 10 Minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No